CLINICAL TRIAL: NCT02624817
Title: Long-term Sulfonylurea Response and Glucose Control After Switching From Insulin in Children With Diabetes Due to KCNJ11 (KIR6.2) Mutations
Brief Title: Long-Term Sulfonylurea Response in KCNJ11 Neonatal Diabetes
Acronym: SuResponsKIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); University of Exeter (Other); Royal Devon and Exeter NHS Foundation Trust (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Hôpital Necker-Enfants Malades (Other); University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 167.06
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Permanent Neonatal Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Permanent Neonatal | interventions — Sulfonylurea Compounds; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: Sulfonylurea (Experimental): Sulfonylurea tablets (glibenclamide, other forms of sulfonylureas) were administered at the time of intervention (before November 1, 2006). The patients have been prospectively followed up. Sulfonylurea dose, insulin requirement, death of all causes, episodes of severe hypoglycemia, ketoacidosis, development of discoloured teeth and diarrhea have been recorded. For a small number of subjects, increment of insulin and C-peptide after either an oral or intravenous glucose load and/or response to glucagon have been tested.
  Interventions: Drug: Sulfonylurea

INTERVENTIONS:
Drug: Sulfonylurea — See Arm description.
  Other Names: Glibenclamide and other forms of sulfonylureas

SUMMARY:
The purpose of this study is to investigate long term response of sulfonylurea and glucose control in children with diabetes due to mutations in KCNJ11 that have been switched from insulin injections to sulfonylurea tablets.

DETAILED DESCRIPTION:
Neonatal diabetes mellitus is a rare, monogenic form of diabetes occurring during the first 6-9 months of life characterized by hyperglycemia requiring exogenous insulin therapy. The estimated incidence is 1 per 12000 newborns. Although homozygous or compound heterozygous mutations in the genes IPF1 or GCK were the first genetic causes of this disease to be identified, activating mutations in the KIR6.2 and sulfonylurea receptor 1 (SUR1) subunits of the pancreatic ATP-sensitive K+ channel, coded for by the genes KCNJ11 and ABCC8, have recently been identified as the major causes of both transient and permanent neonatal diabetes. In the normal pancreatic beta-cell, metabolism results in increased cellular ATP, which binds to KIR6.2. The potassium channel subsequently closes and hence depolarizes the membrane initiating insulin release via increased calcium entry. Conversely, increased cellular ADP acts on SUR1 to open the channel and prevent insulin release. Activating mutations in these channels reduces sensitivity to the inhibitory actions of ATP and increases sensitivity to the stimulatory actions of ADP. This causes the ATP-sensitive K+ channel to remain open, even in the presence of glucose, therefore preventing insulin release. Sulfonylureas act by an ATP-independent mechanism to close these channels even when mutations are present. Sulfonylureas result in insulin release and were therefore immediately considered and showed to be a potential treatment option in neonatal diabetes caused by mutations in these channels. The effective replacement of insulin treatment by high-dose sulfonylureas has been shown to be successful in 90% of patients with Kir6.2 mutations and 85% of patients with SUR1 mutations resulting in improved glycemic control.

This dramatic effect of sulfonylurea is now standard, world-wide treatment in neonatal diabetes due to a mutation in either KCNJ11 or ABCC8. There is, however, far no information on long-term use of sulfonylurea in patients with KCNJ11 or ABCC8 mutations. The investigators have therefore initiated an international, multicenter, prospective study aiming to include some 75 patients aged from 9 years with a genetic diagnosis of diabetes due to a KCNJ11 gene mutation identified by sequencing in Bergen, Norway; Exeter, U.K.; Paris, France or Rome, Italy. Most patients were referred based on membership in the International Society of Pediatric and Adolescent Diabetes. All of the patients attempted transfer from treatment with insulin to a sufficient dose of sulfonylureas. No other selection criteria were applied, and all patients were included when there was outcome data following the attempted transfer. The observation period was at least 9 years after commencing sulfonylureas in all patients. The study is conducted in accordance with the Declaration of Helsinki and informed consent has been obtained from all participating patients, with parental consent given on behalf of children.

ELIGIBILITY:
Inclusion Criteria:

* Permanent diabetes due to a mutation in KCNJ11 (KIR6.2)
* Patients successfully transferred from insulin to sulfonylurea
* Transferred to sulfonylurea treatment before November 1, 2006 (ie 9 years off insulin)
* Willing and able to provide informed consent (parents if younger than 16 years of age)

Exclusion Criteria:

* Permanent diabetes not due to a mutation in KCNJ11 (KIR6.2)
* Patients not successfully transferred from insulin to sulfonylurea
* Transferred to sulfonylurea treatment after November 1, 2006 (ie less than 9 years off insulin)
* Not willing or able to provide informed consent (parents if younger than 16 years of age)

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Sulfonylurea efficacy | Within 13 years from intervention
  Insulin requirement with or without sulfonylurea treatment during the intervention
Metabolic control | Within 13 years from intervention
  Change in HbA1c levels during the intervention

SECONDARY OUTCOMES:
All cause mortality | Within 13 years from intervention
  Death of all causes
Incidence of hypoglycemia | Within 13 years from intervention
  Episodes per year of severe hypoglycemia (ISPAD definitions)
Incidence of ketoacidosis | Within 13 years from intervention
  Episodes per year of severe ketoacidosis (ISPAD definitions)
Development of diarrhea | Within 13 years from intervention
  Chronic diarrhea with no clear cause
Development of discoloured teeth | Within 13 years from intervention
  Discoloured teeth with no clear cause
Insulin secretory response to intravenous glucose | Within 13 years from intervention
  Change in increment of insulin and C-peptide after a standard intravenous glucose tolerance test tested at start of intervention and retested at end of the study
Insulin secretory response to oral glucose | Within 13 years from intervention
  Change in increment of insulin and C-peptide after a standard oral glucose tolerance test tested at start of intervention and retested at end of the study
Sulfonylurea dose | Within 13 years from intervention
  Change in sulfonylurea dose (per kg and day, and absolute dose per day) from start of intervention and up till end of study
Insulin secretory response to a glucagon test | Within 13 years from intervention
  Change in increment of C-peptide and glucose after a standard glucagon test tested at start of intervention and retested at end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pål R Njølstad, MD PhD, Study Director — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Result] Gloyn AL, Pearson ER, Antcliff JF, Proks P, Bruining GJ, Slingerland AS, Howard N, Srinivasan S, Silva JM, Molnes J, Edghill EL, Frayling TM, Temple IK, Mackay D, Shield JP, Sumnik Z, van Rhijn A, Wales JK, Clark P, Gorman S, Aisenberg J, Ellard S, Njolstad PR, Ashcroft FM, Hattersley AT. Activating mutations in the gene encoding the ATP-sensitive potassium-channel subunit Kir6.2 and permanent neonatal diabetes. N Engl J Med. 2004 Apr 29;350(18):1838-49. doi: 10.1056/NEJMoa032922. PMID 15115830
- [Result] Sagen JV, Raeder H, Hathout E, Shehadeh N, Gudmundsson K, Baevre H, Abuelo D, Phornphutkul C, Molnes J, Bell GI, Gloyn AL, Hattersley AT, Molven A, Sovik O, Njolstad PR. Permanent neonatal diabetes due to mutations in KCNJ11 encoding Kir6.2: patient characteristics and initial response to sulfonylurea therapy. Diabetes. 2004 Oct;53(10):2713-8. doi: 10.2337/diabetes.53.10.2713. PMID 15448106
- [Result] Pearson ER, Flechtner I, Njolstad PR, Malecki MT, Flanagan SE, Larkin B, Ashcroft FM, Klimes I, Codner E, Iotova V, Slingerland AS, Shield J, Robert JJ, Holst JJ, Clark PM, Ellard S, Sovik O, Polak M, Hattersley AT; Neonatal Diabetes International Collaborative Group. Switching from insulin to oral sulfonylureas in patients with diabetes due to Kir6.2 mutations. N Engl J Med. 2006 Aug 3;355(5):467-77. doi: 10.1056/NEJMoa061759. PMID 16885550
- [Result] Rafiq M, Flanagan SE, Patch AM, Shields BM, Ellard S, Hattersley AT; Neonatal Diabetes International Collaborative Group. Effective treatment with oral sulfonylureas in patients with diabetes due to sulfonylurea receptor 1 (SUR1) mutations. Diabetes Care. 2008 Feb;31(2):204-9. doi: 10.2337/dc07-1785. Epub 2007 Nov 19. PMID 18025408
- [Result] Stoffers DA, Zinkin NT, Stanojevic V, Clarke WL, Habener JF. Pancreatic agenesis attributable to a single nucleotide deletion in the human IPF1 gene coding sequence. Nat Genet. 1997 Jan;15(1):106-10. doi: 10.1038/ng0197-106. PMID 8988180
- [Result] Njolstad PR, Sovik O, Cuesta-Munoz A, Bjorkhaug L, Massa O, Barbetti F, Undlien DE, Shiota C, Magnuson MA, Molven A, Matschinsky FM, Bell GI. Neonatal diabetes mellitus due to complete glucokinase deficiency. N Engl J Med. 2001 May 24;344(21):1588-92. doi: 10.1056/NEJM200105243442104. No abstract available. PMID 11372010
- [Result] Babenko AP, Polak M, Cave H, Busiah K, Czernichow P, Scharfmann R, Bryan J, Aguilar-Bryan L, Vaxillaire M, Froguel P. Activating mutations in the ABCC8 gene in neonatal diabetes mellitus. N Engl J Med. 2006 Aug 3;355(5):456-66. doi: 10.1056/NEJMoa055068. PMID 16885549
- [Derived] Svalastoga P, Sulen A, Fehn JR, Aukland SM, Irgens H, Sirnes E, Fevang SKE, Valen E, Elgen IB, Njolstad PR. Intellectual Disability in KATP Channel Neonatal Diabetes. Diabetes Care. 2020 Mar;43(3):526-533. doi: 10.2337/dc19-1013. Epub 2020 Jan 13. PMID 31932458
- [Derived] Bowman P, Sulen A, Barbetti F, Beltrand J, Svalastoga P, Codner E, Tessmann EH, Juliusson PB, Skrivarhaug T, Pearson ER, Flanagan SE, Babiker T, Thomas NJ, Shepherd MH, Ellard S, Klimes I, Szopa M, Polak M, Iafusco D, Hattersley AT, Njolstad PR; Neonatal Diabetes International Collaborative Group. Effectiveness and safety of long-term treatment with sulfonylureas in patients with neonatal diabetes due to KCNJ11 mutations: an international cohort study. Lancet Diabetes Endocrinol. 2018 Aug;6(8):637-646. doi: 10.1016/S2213-8587(18)30106-2. Epub 2018 Jun 4. PMID 29880308